CLINICAL TRIAL: NCT03951675
Title: The Burden of Access in Duchenne Muscular Dystrophy in the US. A Qualitative Assessment of the Impact of Access on the Lives of Families Affected by DMD and Their Healthcare Providers.
Brief Title: The Burden of Access in Duchenne Muscular Dystrophy in the US
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Engage Health Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: OCR21561; LHF0001 (Other: WIRB)
Record Dates: First submitted 2019-05-14; First posted 2019-05-15 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals Living with DMD: 90 patients/parents
- Healthcare Providers to Patients with DMD: 40 healthcare providers

SUMMARY:
This study is being conducted to determine if DMD patients / families and healthcare providers experience burdens related to access, and if so, to identify them, and to determine life impacts to the patient, if any, of these burdens. Data from healthcare providers will be collected by an online survey and from patients/families by one on one telephone interview.

DETAILED DESCRIPTION:
Patient/Parent Portion

In this non-interventional study, DMD patients / parents of DMD patients will be interviewed to gather qualitative input, in the patient's voice, regarding challenges associated with access to medications, services and medical equipment, and how these burdens impact quality of life.

Healthcare Provider Portion

In this non-interventional study, healthcare providers who see patients with DMD and who deal with insurance issues on behalf of DMD patients will participate in an online survey designed to determine the burden associated with access to medications, services and medical equipment.

ELIGIBILITY:
Inclusion Criteria:

Patient/Parent interviews

* Patients residing in the US who have been diagnosed with DMD who are age 18 years or older, or the parent / legal guardian of a person of any age who has been diagnosed with DMD,
* Have provide "Proof of DMD" to ensure that they are impacted by the disease,
* Who have provided sufficient information in the RSVP process to determine their functional status; ambulatory, transitional or non-ambulatory,
* State that they are the person who deals with insurance issues for the affected patient and,
* Who are able to understand and consent to participation in the study

Healthcare Provider survey

* Healthcare providers (physicians, nurse practitioners, and physician assistants) currently involved in the care of patients with DMD
* Are currently practicing in the US,
* Who have provided sufficient information in the survey screening to determine that they currently care for DMD patients,
* State that they and/or persons on their staff interface with insurance companies for DMD patients related to access to medications, services and/or medical equipment and,
* Who are able to understand and consent to participation in the study

Exclusion Criteria:

* There are no stated exclusion criteria in this study. Study population must meet all inclusion criteria in order to be deemed eligible to participate.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For Patient/Parent Interviews:
  Patients residing in the US who have been diagnosed with DMD who are age 18 years or older, or the parent / legal guardian of a person of any age who has been diagnosed with DMD
  For Healthcare Provider Survey:
  Healthcare providers (physicians, nurse practitioners, and physician assistants) currently involved in the care of patients with DMD
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-05-28 (Actual)

PRIMARY OUTCOMES:
Burden frequency by functional category | Over 12 months
  The frequency that each burden is mentioned by a patient according to their functional category as measured by the VIGNOS scale. This is the number of times each burden is mentioned by a patient during their interview, assessed by each functional category.

SECONDARY OUTCOMES:
Burden frequency by type of insurance | Over 12 months
  The frequency that each burden is mentioned by a patient according to their insurance coverage. This is the number of times each burden is mentioned by a patient during their interview, assessed by each type of insurance.
Life impact frequency by functional category | Over 12 months
  The frequency that each life impact is mentioned by a patient according to their functional category as measured by the VIGNOS scale. This is the number of times each life impact is mentioned by a patient during their interview, assessed by each functional category.
Life impact frequency by type of insurance | Over 12 months
  The frequency that each life impact is mentioned by a patient according to their insurance coverage. The number of times each life impact is mentioned by a patient during their interview, assessed by each type of insurance.

CONTACTS AND LOCATIONS:
Overall Officials: Kara Godwin, MSN,APRN, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No